CLINICAL TRIAL: NCT02673970
Title: Biomarkers for the Activity of Immune Checkpoint Inhibitor Therapy in Patients With Advanced Melanoma
Acronym: ICIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Bart Neyns, PhD MD Bart Neyns, Universitair Ziekenhuis Brussel
Other Study IDs: 2014-BN-001
Record Dates: First submitted 2016-02-01; First posted 2016-02-04 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Malignant Melanoma
Keywords: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cllection of cell free DNA for mutational analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- observational arm: From start treatment till date of death or date of cure, the patient will be followed for survival and adverse events on pembrolizumab

SUMMARY:
1. Screen and recruitment: patients will be screened based on their prior history and intention to initiate treatment with an immune checkpoint inhibitor.
2. Study phase:

   * Collection of baseline demographic data, prior disease history, nature of ICI therapy, outcome data of ICI therapy (treatment disposition, toxicity, tumor response and survival).
   * Collection of blood samples will be performed every 3 to 4 weeks for the first year on ICI therapy and every 6 to 12 weeks thereafter until the end of ICI therapy, disease progression, death or loss to follow-up. Collection of blood samples will be aligned with the visits necessary for the administration of the ICI therapy.
   * Collection of archival melanoma metastasis tissues will be performed on a continuous basis and be triggered by availability of such tissue following therapeutic resections of melanoma metastases.
3. Follow-up phase

DETAILED DESCRIPTION:
1. Screen and recruitment: patients will be screened based on their prior history and intention to initiate treatment with an immune checkpoint inhibitor. This screening of candidate patients by the investigators will be non-interventional. Patients that are considered eligible candidates will be invited to participate in this study and to Page 3/18 provide written informed consent.
2. Study phase:

   * Collection of baseline demographic data, prior disease history, nature of ICI therapy, outcome data of ICI therapy (treatment disposition, toxicity, tumor response and survival).
   * Collection of blood samples will be performed every 3 to 4 weeks for the first year on ICI therapy and every 6 to 12 weeks thereafter until the end of ICI therapy, disease progression, death or loss to follow-up. Collection of blood samples will be aligned with the visits necessary for the administration of the ICI therapy.
   * Collection of archival melanoma metastasis tissues will be performed on a continuous basis and be triggered by availability of such tissue following therapeutic resections of melanoma metastases.
3. Follow-up phase: patients who stop treatment with the immune checkpoint inhibitor will be followed-up for

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed malignant melanoma;
2. AJCC Stage IIIC or IV melanoma with evaluable disease;
3. Treatment with an immune checkpoint inhibitor;
4. Willing and able to give written informed consent;
5. Accessible for treatment and follow-up;

Exclusion Criteria:

* non

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient with an unresectable stage III or stage IV melanoma treated with pembrolizumab
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-10; Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
explore the value of biomarkers present in blood, and tumor tissue for the purpose of predicting the efficacy of ICI therapy or for the purpose of monitoring the therapeutic effect of ICI therapy | 1year
  explore the value of biomarkers present in blood, and tumor tissue for the purpose of predicting the efficacy of ICI therapy or for the purpose of monitoring the therapeutic effect of ICI therapy

SECONDARY OUTCOMES:
Baseline demographic data, prior disease history, nature of ICI therapy, treatment disposition, adverse events | 1year
  Baseline demographic data, prior disease history, nature of ICI therapy, treatment disposition, adverse events
Tumor response according to the RECISTv1.1 and irRC criteria | 1 year
  Tumor response according to the RECISTv1.1 and irRC criteria
Survival (PFS, and OS) by Kaplan-Meier estimates | 1year
  Survival (PFS, and OS) by Kaplan-Meier estimates
Data collection on the nature and disposition of ICI therapy as well as its efficacy and treatment related adverse events will be collected on a non-interventional basis | 1 year
  Data collection on the nature and disposition of ICI therapy as well as its efficacy and treatment related adverse events will be collected on a non-interventional basis

CONTACTS AND LOCATIONS:
Overall Officials: Bart NEyns, MD; PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (2):
- Belgium (2):
  - UZ Brussel, Jette, Brabant
  - UZ Brussel, Jette, Brussels Capital

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Wilgenhof S, Du Four S, Vandenbroucke F, Everaert H, Salmon I, Lienard D, Marmol VD, Neyns B. Single-center experience with ipilimumab in an expanded access program for patients with pretreated advanced melanoma. J Immunother. 2013 Apr;36(3):215-22. doi: 10.1097/CJI.0b013e31828eed39. PMID 23502769
- [Result] Ribas A, Kefford R, Marshall MA, Punt CJ, Haanen JB, Marmol M, Garbe C, Gogas H, Schachter J, Linette G, Lorigan P, Kendra KL, Maio M, Trefzer U, Smylie M, McArthur GA, Dreno B, Nathan PD, Mackiewicz J, Kirkwood JM, Gomez-Navarro J, Huang B, Pavlov D, Hauschild A. Phase III randomized clinical trial comparing tremelimumab with standard-of-care chemotherapy in patients with advanced melanoma. J Clin Oncol. 2013 Feb 10;31(5):616-22. doi: 10.1200/JCO.2012.44.6112. Epub 2013 Jan 7. PMID 23295794
- [Result] Weber JS, Kudchadkar RR, Yu B, Gallenstein D, Horak CE, Inzunza HD, Zhao X, Martinez AJ, Wang W, Gibney G, Kroeger J, Eysmans C, Sarnaik AA, Chen YA. Safety, efficacy, and biomarkers of nivolumab with vaccine in ipilimumab-refractory or -naive melanoma. J Clin Oncol. 2013 Dec 1;31(34):4311-8. doi: 10.1200/JCO.2013.51.4802. Epub 2013 Oct 21. PMID 24145345
- [Derived] Jansen YJL, Rozeman EA, Mason R, Goldinger SM, Geukes Foppen MH, Hoejberg L, Schmidt H, van Thienen JV, Haanen JBAG, Tiainen L, Svane IM, Makela S, Seremet T, Arance A, Dummer R, Bastholt L, Nyakas M, Straume O, Menzies AM, Long GV, Atkinson V, Blank CU, Neyns B. Discontinuation of anti-PD-1 antibody therapy in the absence of disease progression or treatment limiting toxicity: clinical outcomes in advanced melanoma. Ann Oncol. 2019 Jul 1;30(7):1154-1161. doi: 10.1093/annonc/mdz110. PMID 30923820
- [Derived] de Filette J, Jansen Y, Schreuer M, Everaert H, Velkeniers B, Neyns B, Bravenboer B. Incidence of Thyroid-Related Adverse Events in Melanoma Patients Treated With Pembrolizumab. J Clin Endocrinol Metab. 2016 Nov;101(11):4431-4439. doi: 10.1210/jc.2016-2300. Epub 2016 Aug 29. PMID 27571185